CLINICAL TRIAL: NCT03454750
Title: Radiometabolic Therapy (RMT) With 177Lu PSMA 617 in Advanced Castration Resistant Prostate Cancer (CRPC): Efficacy and Toxicity Evaluation
Brief Title: Radiometabolic Therapy (RMT) With 177Lu PSMA 617 in Advanced Castration Resistant Prostate Cancer (CRPC)
Acronym: LU-PSMA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Istituto Romagnolo per lo Studio dei Tumori Dino Amadori IRST S.r.l. IRCCS (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRST185.03
Record Dates: First submitted 2018-02-27; First posted 2018-03-06 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2025-01

CONDITIONS: Metastatic Castration Resistant Prostate Cancer; 68Ga-PSMA PET/CT Positive
Keywords: Metastatic castration resistant prostate cancer; 68Ga-PSMA PET/CT positive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 177Lu-PSMA (Experimental): 177Lu PSMA
  Interventions: Drug: 177Lu-PSMA

INTERVENTIONS:
Drug: 177Lu-PSMA — 177Lu-PSMA 3.7-5-5 GBq Intravenous Slowly in 15-30 ' Day 1/ every 8-12 weeks Four cycles every 8-12 weeks

SUMMARY:
Radiometabolic Therapy (RMT) with 177Lu PSMA 617 in advanced castration resistant prostate cancer (CRPC): efficacy and toxicity evaluation

DETAILED DESCRIPTION:
Radiometabolic Therapy (RMT) with 177Lu PSMA 617 in advanced castration resistant prostate cancer (CRPC): efficacy and toxicity evaluation. Single-center, prospective, non controlled, open label, phase II trial. The main objective of this study is to evaluate the Disease Control Rate (DCR) and the safety as co-primary objective.

The secondary objectives are: late toxicity, PFS, OS, biochemical response and dosimetry.

ELIGIBILITY:
Inclusion Criteria:

1. Male, Age > 18 years.
2. Patients must have histologically or cytologically confirmation of advanced prostate cancer castration resistant defined according to PCWG3 criteria
3. Measurable disease according to RECIST 1.1. criteria; also patients with bone lesions only could be enrolled
4. Patients with documented disease will be admitted to therapeutic phase only if the diagnostic PET/CT 68Ga-PSMA images demonstrate a significant uptake (tumor to background ratio >2.5) at metastatic tumour site (or in the primary when present, or both)
5. Patients with documented radiological progression (in soft tissue and / or bone) and / or biochemical progression (sequence of 3 PSA rising values from a screening PSA value ≥ 2 ng / ml) according to PCWG3 in pre-study period, refractory or unfit to conventional standard treatments (hormonal or chemotherapeutic treatment such as abiraterone, enzalutamide and docetaxel)
6. Concomitant LHRH analogs assumption is allowed
7. Life expectancy greater than 6 months.
8. ECOG performance status <2
9. Adequate haematological, liver and renal function: haemoglobin >= 9 g/dL, absolute neutrophil count (ANC) >= 1.5 x 109 /L, platelets >= 100 x 109 /L, bilirubin ≤1.5 X upper normal limit (UNL), alanine aminotransferase (ALT) and Aspartate aminotransferase (AST) <2.5 X UNL (< 5 X UNL in presence of liver metastases, creatinine < 2 mg/dL).
10. Participant is willing and able to give informed consent for participation in the study
11. Other known malignant neoplastic diseases in the patient's medical history with a disease-free interval of less than 3 years (except for previously treated basal cell carcinoma).

Exclusion Criteria:

1. Patients treated with chemotherapy and 223Ra radiotherapy within 4 weeks and treated within 2 weeks with palliative radiotherapy.
2. All acute toxic effects of any prior therapy (including surgery, radiation therapy, chemotherapy) must have resolved to a grade ≤ 1 according to National Cancer Institute Common Terminology Criteria for Adverse Events Version 4.03 (CTCAE)
3. ECOG performance status >2
4. Participation in another clinical trial with any investigational agents within 30 days prior to study screening.
5. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
6. Assessed bone marrow invasion > 50%

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 143 (Actual)
Dates: Start 2022-10-25 (Actual); Primary Completion 2024-05-22 (Actual); Study Completion 2024-05-22 (Actual)

PRIMARY OUTCOMES:
Disease Control Rate (DCR ) | up to 36 months
  DCR is defined as the percentage of patients who have achieved complete response, partial response and stable disease lasting for at least 6 months from therapy start. DCR will be evaluated using the new international criteria proposed by the Version 1.1 Response Evaluation Criteria in Solid Tumors (RECIST).
Incidence of Treatment-Emergent Adverse Events | up to 30 days after the last treatment cycle
  The evaluation of the Incidence of Treatment-Emergent Adverse Events starts from the 1st treatment until 30 days after the last treatment cycle; Treatment-Emergent Adverse Events are evaluated according to version 4.03 CTC-AE criteria.

SECONDARY OUTCOMES:
Progression free survival (PFS) | up to 36 months
  PFS is defined as the time from the start treatment date to the date of first observation of documented disease progression or death due to any cause. Patients without tumor progression at the time of analysis will be censored at their last date of tumor evaluation.
Overall survival (OS) | up to 36 months
  Overall survival is defined as the time from the therapy start to the date of death due to any cause or the date of last contact (censored observation) at the date of data cut-off.

CONTACTS AND LOCATIONS:
Overall Officials: Giovanni Paganelli, Study Chair — IRST IRCCS
Locations (1):
- Istituto Scientifico Romagnolo per lo Studio e la Cura dei Tumori (IRST), Meldola, FC, Italy

REFERENCES:
- [Derived] De Giorgi U, Sansovini M, Severi S, Nicolini S, Monti M, Gurioli G, Foca F, Casadei C, Conteduca V, Celli M, Di Iorio V, Calistri D, Matteucci F, von Eyben FE, Attard G, Paganelli G. Circulating androgen receptor gene amplification and resistance to 177Lu-PSMA-617 in metastatic castration-resistant prostate cancer: results of a Phase 2 trial. Br J Cancer. 2021 Oct;125(9):1226-1232. doi: 10.1038/s41416-021-01508-5. Epub 2021 Jul 31. PMID 34333554
- [Derived] Paganelli G, Sarnelli A, Severi S, Sansovini M, Belli ML, Monti M, Foca F, Celli M, Nicolini S, Tardelli E, Marini I, Matteucci F, Giganti M, Di Iorio V, De Giorgi U. Dosimetry and safety of 177Lu PSMA-617 along with polyglutamate parotid gland protector: preliminary results in metastatic castration-resistant prostate cancer patients. Eur J Nucl Med Mol Imaging. 2020 Dec;47(13):3008-3017. doi: 10.1007/s00259-020-04856-1. Epub 2020 May 20. PMID 32430583